CLINICAL TRIAL: NCT01639417
Title: Pilot Functional Imaging Study to Evaluate Mechanisms Underlying Chronic Pain in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Lynn Henry (Other)
Responsible Party: Sponsor-Investigator, Lynn Henry, Principal Investigator, University of Michigan Rogel Cancer Center
Organization: University of Michigan Rogel Cancer Center (Other)
Other Study IDs: UMCC 2011.115; HUM 55687 (Other: HUM 55687); NCT02180594 (obsolete NCT alias)
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Pain; Breast Cancer
MeSH Terms: conditions — Pain; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to better understand why some women with breast cancer develop chronic pain.

DETAILED DESCRIPTION:
Women with breast cancer who either have chronic pain or who do not have chronic pain will be asked to enroll. Those who participate will have pictures taken of their brain using MRI when they are lying still and also when pressure is being applied to their thumbnails. These pictures will be compared to patients without breast cancer who do not have pain and to those who have other types of pain, such as fibromyalgia. By taking and analyzing these pictures the investigators hope to understand more about why breast cancer survivors develop pain after their diagnosis and treatment. In the future the investigators hope to better treat the pain or possibly even prevent the pain from occurring in the first place.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer Survivor with and without chronic pain
* Able to undergo MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer Survivors with and without Chronic Pain
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Determination of differences in pain sensitivity and functional MRI in different groups of patients. | 6 months
  The primary objective of this pilot trial is to determine if there may be differences in mechanical pain sensitivity and functional MRI brain activation patterns in breast cancer survivors with chronic pain as compared to breast cancer patients without chronic pain, to patients with fibromyalgia, or to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Henry, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States